CLINICAL TRIAL: NCT01171235
Title: Study of Previously Collected Blood and Tissue Samples From Patients With Nasopharyngeal Carcinoma,Laryngeal Carcinoma and Hypopharyngeal Carcinoma
Brief Title: Study of Biomarker From Blood and Tissue of Head and Neck Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Southern Medical University, China (Other)
Responsible Party: E.N.T department of Nan Fang Hospital, Nan Fang Medical University, China: National Natural Science Foundation
Other Study IDs: NFYY-H&N-1
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2009-03

CONDITIONS: Laryngeal Neoplasms; Pharyngeal Neoplasms
Keywords: Laryngeal Neoplasms; Pharyngeal Neoplasms
MeSH Terms: conditions — Laryngeal Neoplasms; Pharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and tissue samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study is to find for one or more serum or tissue markers of molecular biology in head and neck cancer patients used for early diagnosis, predicting prognosis and being sensitive to chemotherapy and radiotherapy

DETAILED DESCRIPTION:
Head and neck malignant tumors, especially nasopharyngeal carcinoma in southern China with the high incidence, its incidence, treatment, prognosis or tumor markers in serum has been a hot research with little progress.In our study, we collect NPC-based collection including the blood samples of laryngeal, hypopharyngeal cancer, separating serum and white blood cells stored in -80 degrees，while tissues are frozen in liquid nitrogen and embedded in paraffin。 Patient treatment and prognosis are combined in order to find for markers of molecular biology used for early diagnosis, predicting prognosis and being sensitive to chemotherapy and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* all of nasopharyngeal carcinoma
* hypopharyngeal carcinoma or laryngeal carcinoma visited at ENT department of NanFang hospital

Exclusion Criteria:

* all of above patients whose anticipated survival duration were less than 6 months

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all of nasopharyngeal carcinoma, hypopharyngeal carcinoma or laryngeal carcinoma visited at ENT department of NanFang hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ping Xiang Li, doctor, Study Director — E.N.T department of NanFang hospital

REFERENCES:
- [Derived] Yu BL, Peng XH, Zhao FP, Liu X, Lu J, Wang L, Li G, Chen HH, Li XP. MicroRNA-378 functions as an onco-miR in nasopharyngeal carcinoma by repressing TOB2 expression. Int J Oncol. 2014 Apr;44(4):1215-22. doi: 10.3892/ijo.2014.2283. Epub 2014 Jan 28. PMID 24481647